CLINICAL TRIAL: NCT02532010
Title: Induction Therapy With Pacritinib Combined With Decitabine or Cytarabine in Older Patients With Acute Myeloid Leukemia (AML)
Brief Title: Pacritinib Combined With Decitabine or Cytarabine in Older Patients With AML
Acronym: Pacritinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was put on clinical hold by the sponsor since Feb 9th 2016, and was later decided not to re-open due to financial constraints.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1403014921
Record Dates: First submitted 2015-08-06; First posted 2015-08-25 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Decitabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Pacritinib and Decitabine (Active Comparator): Arm A: Each cycle: Decitabine 20mg/m2 intravenous daily for 10 days combined with ongoing pacritinib 200 mg twice daily.
  Interventions: Drug: Pacritinib; Drug: Decitabine
- Arm B: Pacritinib and Cytarabine (Active Comparator): Arm B: Each cycle: Cytarabine 20mg subcutaneous twice daily for 10 days combined with ongoing pacritinib 200mg twice daily.
  Interventions: Drug: Pacritinib; Drug: Cytarabine

INTERVENTIONS:
Drug: Pacritinib — Pacritinib is a novel Janus kinase 2-fms-like receptor tyrosine kinase 3 (JAK2-FLT3) inhibitor that has shown promising antitumor activity. Pacritinib is a potent inhibitor of JAK2 and FLT3 kinase activities (50% inhibitory concentration (IC50) = 23 nanomolar (nM)and 22 nM, respectively). The drug also inhibits cellular proliferation in human leukemia and lymphoma cell lines selected for their dependence on either of the target kinases. Consistent with these activities, exposure to pacritinib resulted in the reduction of phos-JAK2, phos-STAT3 or phos-STAT5 in the relevant cell lines. Unlike some JAK2 inhibitors, pacritinib does not inhibit Janus kinase 1 (JAK1).
  Other Names: SB1518
Drug: Decitabine — Commercial drug: For each cycle Decitabine 20mg/m2 intravenous daily for 10 days combined with ongoing pacritinib 200 mg twice daily.
  Other Names: Dacogen
  Arms: Arm A: Pacritinib and Decitabine
Drug: Cytarabine — Commercial drug: For each cycle Cytarabine 20mg subcutaneous twice daily for 10 days combined with ongoing pacritinib 200mg twice daily.
  Other Names: Cytosar-U, Tarabine PFS, Cytosar
  Arms: Arm B: Pacritinib and Cytarabine

SUMMARY:
The purpose of this study is to see if a medicine called pacritinib is both safe and effective as a study intervention for patients with AML in combination with either decitabine or cytarabine. Pacritinib is an experimental drug that is being studied to treat acute myeloid leukemia (AML). Decitabine and cytarabine are both FDA approved drugs that are used in treatment of AML. Pacritinib is being tested in clinical trials and has not been submitted to the U.S. Food and Drug Administration (FDA) for approval for any indications. Pacritinib is a drug that is designed to slow down the growth of leukemic cells.

DETAILED DESCRIPTION:
This is a single-center, open label, two-arm phase II study of clinical activity of pacritinib in older patients newly diagnosed with AML combined with either decitabine or cytarabine. In this study, approximately 61 patients will be enrolled at the Weill Cornell Medical College. Arm A consists of pacritinib and decitabine and will enroll 31 subjects, and Arm B consists of pacritinib and cytarabine and will enroll 30 subjects. Arm A and B will enroll sequentially. The dose of pacritinib will be 200mg twice a day continuously.

Arm A: Each cycle: Decitabine 20mg/m2 intravenous daily for 10 days combined with ongoing pacritinib 200 mg twice daily.

Arm B: Each cycle: Cytarabine 20mg subcutaneous twice daily for 10 days combined with ongoing pacritinib 200mg twice daily.

Treatment may be given on an outpatient basis if hospitalization is not otherwise required. Every effort should be made to give decitabine or cytarabine consecutively for 10 days; however if interruption is needed, discussion will be held with the medical monitor and the investigator.

The first day of a cycle will be defined as the day on which decitabine or cytarabine is started. First treatment will take place on Cycle 1, day 1. Hydroxyurea may be used at the investigator's discretion for the first 28 days on Cycle 1 to maintain white blood cell count (WBC) <30,000/µl. Bone marrow biopsy and aspiration will be performed between days 22-56 of each cycle and the subsequent treatment cycle will be started between days 22-56, at the investigator's discretion. Ideally, cycles will be administered at 28-day intervals, but treatment delays of decitabine or cytarabine up to 56 days will be permitted to allow resolution of non-hematologic and non-disease-related hematologic toxicities. Granulocyte-stimulating cytokine support will be permitted at the investigator's discretion in the event of neutropenic fever/sepsis as per American Society of Clinical Oncology (ASCO) guidelines.16 Bone marrow aspiration and biopsy will be performed within 5 days of peripheral blood count recovery to an absolute neutrophil count (ANC) ≥ 1000/µL and platelets ≥ 100,000/µL without transfusions, or day 28 whichever comes first. If the peripheral blood absolute blast count is ≥ 5000/µL on day 21 of the first cycle, the second cycle may be administered immediately after bone marrow aspiration and biopsy.

Each arm will enroll in a Simon's two-stage design as described in Section 8. In Arm A, 16 subjects will initially be entered into the study, and if 6 or fewer respond, then Arm A will be terminated early and study will proceed to Arm B. In Arm B, 15 subjects will initially be entered into the study, and if 2 or fewer respond, the study will be terminated early.

Duration of study therapy Patients will receive a minimum of 4 cycles of treatment unless there is evidence of unacceptable regimen-related toxicity or unequivocal disease progression for which the investigator is specifically recommending alternative therapy. Pacritinib will continue throughout the study.

Arm A:

Patients who achieve Complete Remission (CR), Complete Remission with incomplete platelet recovery (CRp), or complete remission with incomplete blood count recovery (CRi) will receive subsequent cycles of decitabine on a monthly basis with decitabine 20mg/m2 IV daily for 5 days with pacritinib. Patients who do not achieve complete remission, but who are responding to treatment (partial response, hematologic response, or clinical benefit as determined by the investigator) will receive four 10-day cycles of decitabine with pacritinib as indicated in the study design, followed by monthly maintenance cycles of decitabine 20mg/m2 IV daily for 5 days + daily pacritinib. The maintenance cycles will continue indefinitely until relapse or toxicity. Patients may be taken off study for allogeneic stem cell transplantation at the discretion of the investigator.

Arm B:

Patients will continue cytarabine 20mg subcutaneous twice daily for 10 days combined with pacritinib for up to 4 cycles to achieve CR, CRp, or CRi. Those patients who achieve CR, CRp, or CRi after 4 cycles may continue to receive monthly maintenance of cytarabine 20mg subcutaneous twice daily for 10 days with pacritinib. The maintenance cycles will continue indefinitely until relapse or toxicity. Patients may be taken off study for allogeneic stem cell transplantation at the discretion of the investigator.

Screening (Study Day -14 to Day 1) Initiate and complete screening activities within 14 days before Cycle 1, Day 1 treatment.

Treatment (Cycle 1, Day 1 through End-of-Treatment Visit) This period begins on the day the patient first receives treatment and ends at the End-of-Treatment Visit.

Follow-up After completion of the End-of-Treatment Visit, all patients are followed up for 30 days and followed every three months for survival and disease status.

Clinical Study Endpoints The Primary objective of the study is to evaluate the safety and efficacy of pacritinib combined with decitabine or cytarabine in newly diagnosed older (≥65 years old) patients with AML. The primary endpoint of this study will be complete remission according to the International Working Group (IWG) criteria.

The following secondary endpoints will be evaluated:

* Overall Survival (OS)
* Overall remission (OS) rate, defined as CR + CRp + Cri + Partial Remission (PR) based on IWG response criteria
* Relapse-free Survival (RFS)
* Event-free Survival (EFS)
* Time to Complete Response (TTCR)
* Remission Duration

DISCUSSION OF STUDY DESIGN

Prognosis for older patients with AML is poor, with median survival of only 9-12 months. Older patients are often not candidates for intensive chemotherapy or allogeneic stem cell transplantation. Decitabine and low-dose cytarabine are frequently used for upfront treatment of older AML patients, however CR rates are 40-50% with decitabine and 18% with cytarabine. Pacritinib is a potent tyrosine kinase inhibitor of FLT3 and Janus Kinase 3 (JAK3) tyrosine kinases. The objective of the proposed clinical trial is to evaluate the efficacy, safety, and feasibility of pacritinib combined with decitabine or cytarabine in newly diagnosed older AML patients. The primary endpoint will be increase in complete remission.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has unequivocal pathologic diagnosis of AML (≥ 20% blasts in the bone marrow based on World Health Organization (WHO) criteria), excluding acute promyelocytic leukemia t(15;17)(q22;q12); Promyelocytic leukemia gene (PML)- retinoic acid receptor alpha (RARA)
2. Age ≥ 65 years old
3. No prior treatment for AML except:

   * Emergency leukapheresis
   * Emergency treatment for hyperleukocytosis with hydroxyurea
   * Cranial radiotherapy (RT) for Central Nervous System (CNS) leukostasis (one dose only)
   * Growth factor/cytokine support
4. AML patients with therapy-related myeloid neoplasms are eligible if they have not received radiation therapy or chemotherapy (not including hormonal therapy) for their primary malignancy or disorder for ≥ 6 months. Hydroxyurea may be used at the investigator's discretion up to the first 28 days on Cycle 1 to maintain WBC <30,000/µl.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
6. Subjects must have adequate hepatic and renal function
7. Female subject of child-bearing potential and male subjects with female partners of reproductive potential must use acceptable contraceptive methods
8. Able to understand and to provide written informed consent
9. Able to comply with all study procedures during the study including all visits and tests
10. Willing to adhere to the prohibitions and restrictions specified in this protocol
11. Patient must sign an informed consent form (ICF)

Exclusion Criteria:

1. Prior treatment with decitabine
2. Prior treatment with cytarabine
3. Prior treatment with pacritinib
4. Presence of serious illness, medical condition, or other medical history, involving the heart, kidney, liver, or other organ system, including abnormal laboratory parameters, which, in the opinion of the Investigator, would be likely to interfere with a subject's participation in the study or with the interpretation of the results.
5. Active, uncontrolled, clinically significant infection(s)
6. Have other active malignancies (excluding other myeloid hematologic malignancies) or other malignancies within 12 months before enrollment, except curatively treated non-melanoma skin cancer, cervical intraepithelial neoplasia, organ-confined or treated non-metastatic prostate cancer with negative prostate-specific antigen, in situ breast carcinoma after complete surgical resection, or superficial transitional cell bladder carcinoma
7. Are receiving any other investigational therapy or protocol-prohibited therapy
8. Any prior or co-existing medical condition that in the Investigator's judgment will substantially increase the risk associated with the subject's participation in the study
9. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures
10. Any gastrointestinal (GI) or metabolic condition that could interfere with absorption of oral medication
11. Inflammatory or chronic functional bowel disorder, such as Crohn's disease, inflammatory bowel disease, chronic diarrhea
12. Clinically symptomatic and uncontrolled cardiovascular disease
13. History of any of the following within 6 months: myocardial infarction, severe/unstable angina, or symptomatic congestive heart failure
14. New York Heart Association Class III or IV congestive heart failure
15. Patients with National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) grade 2 cardiac arrhythmias may be considered for inclusion with the approval of the investigator if the arrhythmias are stable, asymptomatic and unlikely to affect patient safety. Patients will be excluded if they have ongoing cardiac dysrhythmias of CTCAE grade 3, corrected QT interval (QTc) prolongation >450 ms by Fridericia method, or other factors that increase the risk for QT prolongation (eg, heart failure, hypokalemia [defined as serum potassium < 3.0 milliequivalent (mEq/L) that is persistent and refractory to correction], or family history of long QT interval syndrome).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2016-02-09 (Actual); Study Completion 2017-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SangMin Lee, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
data will be shared with the sponsor

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Pacritinib and Decitiabine: Arm A: Each cycle: Decitabine 20mg/m2 intravenous daily for 10 days combined with ongoing pacritinib 200 mg twice daily.
  Pacritinib: Pacritinib is a novel Janus kinase 2-fms-like receptor tyrosine kinase 3 (JAK2-FLT3) inhibitor that has shown promising antitumor activity. Pacritinib is a potent inhibitor of JAK2 and FLT3 kinase activities (50% inhibitory concentration (IC50) = 23 nM and 22 nM, respectively). The drug also inhibits cellular proliferation in human leukemia and lymphoma cell lines selected for their dependence on either of the target kinases. Consistent with these activities, exposure to pacritinib resulted in the reduction of phos-JAK2, phos-STAT3 or phos-STAT5 in the relevant cell lines. Unlike some JAK2 inhibitors, pacritinib does not inhibit JAK1.
  Decitabine: Commercial drug: For each cycle Decitabine 20mg/m2 intravenous daily for 10 days combined with ongoing pacritinib 200 mg twice daily.
- Arm B: Pacritinib and Cytarabine: Arm B: Each cycle: Cytarabine 20mg subcutaneous twice daily for 10 days combined with ongoing pacritinib 200mg twice daily.
  Pacritinib: Pacritinib is a novel Janus kinase 2-fms-like receptor tyrosine kinase 3 (JAK2-FLT3) inhibitor that has shown promising antitumor activity. Pacritinib is a potent inhibitor of JAK2 and FLT3 kinase activities (50% inhibitory concentration (IC50) = 23 nM and 22 nM, respectively). The drug also inhibits cellular proliferation in human leukemia and lymphoma cell lines selected for their dependence on either of the target kinases. Consistent with these activities, exposure to pacritinib resulted in the reduction of phos-JAK2, phos-STAT3 or phos-STAT5 in the relevant cell lines. Unlike some JAK2 inhibitors, pacritinib does not inhibit JAK1.
  Cytarabine: Commercial drug: For each cycle Cytarabine 20mg subcutaneous twice daily for 10 days combined with ongoing pacritinib 200mg twice daily.
Period: Overall Study
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine
Started | 9 | 4
Completed | 0 | 0
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 9 | 4 | 13
Age, Continuous [Median (Full Range); unit: years] | 76 [70 to 84] | 73 [68 to 75] | 75 [68 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 2 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate
Description: Complete remission rate is defined as number of subjects with complete remission according to the IWG criteria, which is defined by presence of <5 percent of blasts in the bone marrow, absence of blasts with Auer rods, absence of extramedullary disease, absolute neutrophil count >1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100,000/µL); independence of red cell transfusions.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine
Number analyzed (Participants) | 9 | 4
Participants | 0 | 0

2. Secondary Outcome: Overall Survival
Description: Survival following treatment to the date of death
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine
Number analyzed (Participants) | 9 | 4
Participants | 3 | 3

3. Secondary Outcome: Overall Remission Rate
Description: Overall remission rate is defined as number of subjects with complete remission (CR), Complete Remission with incomplete platelet recovery (CRp), Complete Remission with Incomplete Blood Count Recovery (CRi), Partial Remission (PR) according to the IWG criteria. CRi is defined as All CR criteria except for residual neutropenia (<1.0 x 109/L (1000/µL)) or thrombocytopenia (<100 x 109/L (100,000/µL)), PR is defined as relevant in the setting of phase I and II clinical trials only; all hematologic criteria of CR; decrease of bone marrow blast percentage to 5 to 25 percent; and decrease of pretreatment bone marrow blast percentage by at least 50 percent.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine
Number analyzed (Participants) | 9 | 4
Participants | 0 | 0

4. Secondary Outcome: Relapse-free Survival
Description: Time from complete remission documentation to either AML relapse or death from any cause.
Time Frame: From date of complete remission until either AML relapse or death from any cause, whichever came first, assessed throughout the study period up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine
Number analyzed (Participants) | 9 | 4
months | NA [NA to NA] — No patients achieved complete remission | NA [NA to NA] — No patients achieved complete remission

5. Secondary Outcome: Event-free Survival
Description: Time from entry on study until time at which there is treatment failure, AML relapse, or death from any cause
Time Frame: Time from entry on study until time at which there is treatment failure, AML relapse, or death from any cause, assessed throughout the study period up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine
Number analyzed (Participants) | 9 | 4
months | 2.5 [2 to 4] | 3 [1 to 5]

6. Secondary Outcome: Time to Complete Response
Description: Time from entry on study until documentation of complete remission (CR)
Time Frame: From entry on study until complete remission, assessed throughout the study period up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine
Number analyzed (Participants) | 9 | 4
months | NA [NA to NA] — No patients achieved complete remission | NA [NA to NA] — No patients achieved complete remission

7. Secondary Outcome: Remission Duration
Description: Time from CR documentation to AML relapse
Time Frame: time from complete remission to AML relapse, assessed throughout the study period up to 2 years.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine
Number analyzed (Participants) | 9 | 4
months | NA [NA to NA] — No patients achieved complete remission | NA [NA to NA] — No patients achieved complete remission

ADVERSE EVENTS:
Time Frame: 2 years, 4 months
Arm/Group | Arm A: Pacritinib and Decitiabine | Arm B: Pacritinib and Cytarabine
All-Cause Mortality (participants affected / at risk) | 9/9 | 4/4
Serious Adverse Events (participants affected / at risk) | 9/9 | 4/4
Other Adverse Events (participants affected / at risk) | 9/9 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pacritinib and Decitiabine (N=9) | Arm B: Pacritinib and Cytarabine (N=4)
Dizziness and right shoulder pain (Nervous system disorders) | 0 (0) | 1 (1)
fever (General disorders) | 0 (0) | 1 (1)
presyncope (Nervous system disorders) | 0 (0) | 1 (1)
neutropenic fever (Blood and lymphatic system disorders) | 2 (3) | 2 (4)
failure to thrive (General disorders) | 1 (1) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 2 (2) | 0 (0)
dehydration/diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 0 (0)
fall (General disorders) | 1 (1) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
oral ulceration (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pacritinib and Decitiabine (N=9) | Arm B: Pacritinib and Cytarabine (N=4)
nausea (Nervous system disorders) | 7 (7) | 4 (6)
anorexia (General disorders) | 3 (3) | 2 (4)
dizziness (Nervous system disorders) | 4 (4) | 3 (4)
vomiting (Gastrointestinal disorders) | 4 (4) | 2 (5)
fatigue (General disorders) | 8 (8) | 2 (3)
insomnia (Psychiatric disorders) | 6 (6) | 1 (1)
constipation (Gastrointestinal disorders) | 7 (7) | 2 (2)
bleeding gums (General disorders) | 1 (1) | 1 (1)
dry mouth (General disorders) | 4 (4) | 1 (1)
fall (General disorders) | 6 (6) | 4 (4)
ecchymosis on buttocks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (3)
bacteremia (Infections and infestations) | 1 (1) | 2 (2)
non-obstructing renal calculi/hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
mucositis (Gastrointestinal disorders) | 3 (3) | 3 (3)
chest pain (Cardiac disorders) | 4 (4) | 2 (2)
hypertension (Vascular disorders) | 0 (0) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
creatinine increased (Investigations) | 2 (2) | 1 (1)
presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (8) | 3 (4)
Chills (General disorders) | 4 (4) | 3 (3)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Fever (General disorders) | 1 (1) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
hypovolemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0)
bilateral leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
anxiety (Nervous system disorders) | 3 (3) | 0 (0)
LE edema (General disorders) | 5 (5) | 3 (3)
coagulpathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
loss of appetite (General disorders) | 2 (2) | 2 (2)
maculo-papular rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
hallucinations (Nervous system disorders) | 2 (2) | 0 (0)
oral sore (General disorders) | 1 (1) | 0 (0)
pruitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hemorraghic bullae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
nocturia (Renal and urinary disorders) | 1 (1) | 1 (1)
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
drug rash (Investigations) | 2 (2) | 0 (0)
hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
external hemorrhoids (Renal and urinary disorders) | 2 (2) | 0 (0)
tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
rigors (General disorders) | 2 (2) | 1 (1)
Asteatotic eczema and xerosis lower legs and elbows (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
pruitic groin (Infections and infestations) | 1 (1) | 0 (0)
non-specific body pain (General disorders) | 1 (1) | 0 (0)
pyuria (Infections and infestations) | 1 (1) | 0 (0)
sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
rash on trunk/legs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
increased urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
oral thrush (Infections and infestations) | 1 (1) | 0 (0)
great toe pain (General disorders) | 1 (1) | 0 (0)
tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
dysuria (Infections and infestations) | 1 (1) | 0 (0)
congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
NSVT (Cardiac disorders) | 1 (1) | 0 (0)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
urinary distention (Renal and urinary disorders) | 1 (1) | 0 (0)
sacral pressure ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
temporal wasting (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
right eye conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
hypotension (Vascular disorders) | 5 (5) | 1 (1)
hypernatremia (Investigations) | 2 (2) | 0 (0)
confusion (Psychiatric disorders) | 1 (1) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0)
hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
generalized weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
nare lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
internal hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
mucocutaneous pain (Infections and infestations) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 2 (2) | 0 (0)
R shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
loose stool (Gastrointestinal disorders) | 1 (1) | 2 (2)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
delirium (Psychiatric disorders) | 1 (1) | 0 (0)
right chest pain (General disorders) | 1 (1) | 0 (0)
left chest pain (General disorders) | 1 (1) | 0 (0)
troponin I increased (Investigations) | 1 (1) | 0 (0)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
VRE bacteremia (Infections and infestations) | 2 (2) | 0 (0)
pitting edema (General disorders) | 1 (1) | 1 (1)
intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
toenail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
tremors (Nervous system disorders) | 1 (1) | 0 (0)
bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
stomach burning (Gastrointestinal disorders) | 1 (1) | 0 (0)
oral herpes sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dry nasal passages (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
L eye ecchymoses (Eye disorders) | 1 (1) | 0 (0)
intermittent swelling in feet (General disorders) | 1 (1) | 0 (0)
polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
petechiae on extremities (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
b/l LE weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
b/l feet purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
blanching erythmatous rash on arm and back (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
eye floaters (Eye disorders) | 0 (0) | 1 (1)
R wrist hematoma (Vascular disorders) | 0 (0) | 1 (1)
hypophosphatemia (Investigations) | 3 (3) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pleural effusions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
septic shock (Infections and infestations) | 0 (0) | 1 (1)
elevated lactate (Investigations) | 0 (0) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
decreased appetite (Gastrointestinal disorders) | 2 (2) | 0 (0)
C. diff colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
polymicrobial sepsis (Infections and infestations) | 1 (1) | 0 (0)
gas pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
altered mental status (Psychiatric disorders) | 1 (1) | 0 (0)
oliguyric AKI (Renal and urinary disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0)
hypoalbuminemia (Investigations) | 2 (3) | 0 (0)
stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0)
rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
rash on arms/legs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
oral ulceration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
sore on tongue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
numbness in feet (Nervous system disorders) | 2 (2) | 0 (0)
avulsed toenail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dry right sole of foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
R sided dental pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypocalcemia (Investigations) | 1 (1) | 1 (1)
edema (General disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
fatigue upon exertion (General disorders) | 0 (0) | 1 (1)
atypical pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sweats (General disorders) | 0 (0) | 1 (1)
lung infection (Infections and infestations) | 0 (0) | 1 (1)
diffuse rash on trunk (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
erythematous lesion on L forearm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
lightheadedness (Nervous system disorders) | 1 (3) | 1 (1)
hives following platelet transfusion (General disorders) | 0 (0) | 1 (1)
hyperglycemia (Investigations) | 1 (1) | 0 (0)
increased LDH (Investigations) | 1 (1) | 0 (0)
forceful urination (Renal and urinary disorders) | 1 (1) | 0 (0)
prolonged QTc interval (Cardiac disorders) | 1 (1) | 0 (0)
malaise (General disorders) | 1 (1) | 0 (0)
intermittent chest palpitations (Cardiac disorders) | 1 (1) | 0 (0)
night sweats (General disorders) | 2 (2) | 0 (0)
R hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
numbness in fingers (Nervous system disorders) | 1 (1) | 0 (0)
body aches (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
b/l rash on groin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RLQ papular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No